CLINICAL TRIAL: NCT03437694
Title: Assessing the Impact of Providing Pharmacists With Medical Records in a Patient-Centered, Community Pharmacy-Based, HIV Care Model
Brief Title: Impact of Providing Medical Records in a Patient-Centered, Community Pharmacy Based, HIV Care Model (HIV-MOI)
Acronym: HIV-MOI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and funding challenges
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: University of California, San Francisco (Other); University of Minnesota (Other); Walgreens Boots Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: U54Proj2
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Diabetes Mellitus, Type 2; Hypertension
Keywords: HIV; AIDS; Diabetes Melllitus, Type 2; Hypertension; Pharmacist; Medication optimization; Medication Therapy Management; MTM
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diabetes Mellitus, Type 2; Hypertension | interventions — Medication Therapy Management

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either the intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication Optimization Intervention (Experimental): This group will represent those participants whose medical records have been provided to the pharmacist.
  Interventions: Other: Medication optimization intervention
- Medication Optimization Control (Active Comparator): This group will represent those participants whose medical records have not been provided to the pharmacist.
  Interventions: Other: Medication optimization intervention

INTERVENTIONS:
Other: Medication optimization intervention — Pharmacists will engage participants in medication therapy management either with access to the medical records (intervention) or without access (control).
  Other Names: medication therapy management

SUMMARY:
This is a clinical trial. The purpose of this clinical trial is to see if study participants have better health outcomes if their pharmacist has access to their medical records. The study will take place primarily in Fort Worth and Dallas, Texas. The trial will enroll adult, African-Americans with HIV. Study participants must also have either diabetes, high blood pressure or they may have both. Study participants will agree to have their medical records from all of their health providers released to UNTHSC. UNTHSC will provide the study pharmacist the medical records for half of the participants. Using the medical records, the study pharmacist will provide 'enhanced' patient counseling services to half of the participants. This enhanced service is called 'medication optimization'. For half of the participants that the study pharmacist does not see the medical records, they will receive usual and customary patient counseling. Not seeing the medical records is considered standard of care. In both groups, the counseling frequency will be based on the participant's needs but the study pharmacist will contact every participant to check on them at least every 90 days. These visits will happen for 2 years. The two groups will be compared to see if those participants having medical information supported medication optimization have better health than those getting routine, the standard of care medication optimization.

DETAILED DESCRIPTION:
This study examines HIV medication optimization (HIV-MOI) in a prospective, randomized (1:1 HIV-MOI: standard of care), clinical trial, comparing disease-specific clinical and humanistic outcomes in up to 200 adult African-Americans with HIV (1:1 men: women) and either diabetes mellitus type 2 (DM) and/or hypertension (HTN). Data will be collected from individual participants for a 2 year period. Once properly screened, consented and enrolled, medical records from participant's medical provider(s) will be obtained. Upon receipt of the medical records, research team personnel (working closely with the project biostatistician) will provide medical information only for those participants randomized to receive HIV-MOI to the study pharmacist. The study pharmacist then assesses the information to determine the clinical effectiveness and appropriateness of the current medical plan's medications. Upon completion, the study pharmacist will develop a prioritized medication problem list, create a plan, discuss/collaborate with the medical provider/healthcare team member as needed and then conduct the initial HIV-MOI visit with the patient. At the initial visit, an individualized care plan would be finalized with study participant input. Also at the initial HIV-MOI visit, the patient should receive an accurate (and reconciled with medical providers) personal medication record (PMR). Participants should also receive an individualized care plan called a medication action plan (MAP). The MAP can include non-pharmacological instructions and education. This may be guided in part by qualitative survey data obtained as part of the study visit. Follow-up visits will occur (ideally) not less than quarterly. Follow-up visits may occur face-to-face or using telecommunication methods.

The study pharmacist will only be provided the medical information for the intervention group. Standard of care for pharmacists is not having access to medical information when providing HIV-MOI. Extracted data and study obtained data will be entered into the study database for analyses.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* African-American
* HIV positive
* At least one of the following: hypertension or diabetes type 2

Exclusion Criteria:

* Pregnant (at screening, may enroll 6 months post-delivery)
* Have a life expectancy < 2 years
* Refusal to provide medical record release

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal K Hodge, PharmD, Principal Investigator — UNTHSC
Locations (2):
- United States (2):
  - Crystal Hodge, Fort Worth, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: The study coordinator would request medical records for study participants in the intervention arm in compliance with Texas state laws and aggregate pertinent information (ex: labs) into a prespecified case report form. The case report form was provided to the study pharmacist conducting MTM during study visits with study participants.
- Control Arm: The study pharmacist conducted MTM with the study participants per standard of care (i.e. additional medical records information was not provided).
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 64 | 65
Completed | 25 (Completed all 9 study visits) | 26 (Completed all 9 study visits)
Not Completed | 39 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at time of study enrollment expressed as years
  years | 54.01 (10.6) | 52.38 (10.96) | 53.19 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 37 | 41 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-identification as African American or Black was an inclusion criteria for this study. Other race and ethnicity data was not collected.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 64 | 65 | 129
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
HIV Viral Load [Count of Participants; unit: Participants]
  VL < LLOQ | 18 | 29 | 47
  Detectable VL | 46 | 36 | 82
Comorbidities [Count of Participants; unit: Participants]
  Hypertension | 43 | 34 | 77
  Diabetes mellitus | 21 | 31 | 52

OUTCOME MEASURES:

1. Primary Outcome: Average A1c
Description: The average A1c in study participants with Diabetes mellitus at the end of their study participation
Time Frame: Through study completion, up to 3 years
Population: Only study participants with Diabetes mellitus
Measure: Mean (Standard Deviation); unit: Average A1c (% glyosylated hemoglobin)
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 21 | 31
Average A1c (% glyosylated hemoglobin) | 7.45 (1.84) | 6.66 (2.26)

2. Primary Outcome: Average Systolic Blood Pressure
Description: The average SBP in study participants with hypertension at the end of their study participation
Time Frame: Through study completion, up to 3 years
Population: Only study participants with hypertension
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 43 | 34
mmHg | 134.6 (13.1) | 129.2 (14.9)

ADVERSE EVENTS:
Time Frame: Through study completion, up to 3 years
Description: Serious adverse events included any hospitalization for any cause including scheduled procedures or unrelated hospitalizations. Other adverse events were not monitored or assessed
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 1/64 | 1/65
Serious Adverse Events (participants affected / at risk) | 8/64 | 9/65
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=64) | Control Arm (N=65)
Hospitalization due to procedure or surgery (Surgical and medical procedures) | 1 (1) | 2 (2)
Hospitalization unscheduled (General disorders) | 7 (7) | 5 (5) — Causes varied from infection to fall or unknown. None were deemed to be associated with the study.
ED visit (General disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Challenges with recruitment during the COVID-19 pandemic limited study participant enrollment within the grant period. Due to funding and enrollment constraints, the study was terminated before all study participants were able to complete all expected study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT03437694/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03437694/ICF_001.pdf